CLINICAL TRIAL: NCT02116582
Title: A Multi-center, Single Arm Study of Enzalutamide in Patients With Progressive Metastatic Castration-Resistant Prostate Cancer Previously Treated With Abiraterone Acetate
Brief Title: A Study to Evaluate Enzalutamide After Abiraterone in Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0410; 2013-002271-17 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: MDV3100; Xtandi; Abiraterone; Metastatic Castration-Resistant Prostate Cancer; Enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enzalutamide (Experimental): Participants received 160 mg of enzalutamide orally once daily until they experienced an adverse event, disease progression, started new anti-cancer therapy, withdrew consent, or other protocol-specified criteria.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Participants received 160 mg of enzalutamide (soft capsules) orally once daily.
  Other Names: MDV3100; Xtandi

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of enzalutamide treatment in patients with progressive metastatic castration-resistant prostate cancer previously treated with abiraterone acetate.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed adenocarcinoma of the prostate without neuro-endocrine differentiation or small cell features.
* Subject has metastatic disease documented by bone scan or by soft tissue disease observed by Computed Tomography/Magnetic Resonance Imaging (CT/MRI) at screening, or within ≤30 days prior to Day 1.
* In the setting of castrate levels of testosterone ≤1.7 nmol/L (or ≤50 ng/dL), subject has progressive disease at study entry defined as PSA rise determined by a minimum of 2 rising PSA levels with an interval of ≥ 1 week between each assessment. The PSA value at the screening visit should be ≥ 2 ng/mL WITH or WITHOUT:

  * Soft tissue disease progression defined by Response Evaluation Criteria In Solid Tumors (RECIST 1.1) at screening, or within ≤30 days prior to Day 1. Measurable disease is not required for entry. Lymph nodes ≥ 2 cm are considered measurable disease (Prostate Cancer Clinical Trials Working Group (PCWG2)).
  * Bone disease progression defined by at least 2 new lesions on bone scan at screening, or within ≤30 days prior to Day 1.
* Subject must have received a minimum of 24 weeks of treatment with abiraterone acetate within its approved label indication and has discontinued use at least 4 weeks prior to start of study drug at Day 1.
* If the subject has received previous treatment with chemotherapy for prostate cancer, this must be limited to no more than one prior line of docetaxel, and must have been used prior to abiraterone acetate therapy.
* Subject receives and will continue to receive ongoing androgen deprivation with Luteinizing-hormone-releasing hormone (LHRH) analogue therapy throughout the course of the study or has had a bilateral orchiectomy.
* Subject is asymptomatic or mildly symptomatic from prostate cancer:

  * The score on Brief Pain Inventory - Short Form (BPI-SF) Question #3 must be < 4.
  * No use of opiate analgesics for prostate cancer-related pain currently or anytime within 4 weeks prior to screening.

Exclusion Criteria:

* Subject has prior use of ketoconazole for the treatment of prostate cancer.
* Subject has prior use of cabazitaxel.
* Subject has prior use of enzalutamide.
* Subject has received ANY anti-neoplastic therapy (including antiandrogens and chemotherapy) following abiraterone acetate discontinuation and prior to start of study drug at Day 1.
* Subject has a known or suspected hypersensitivity to enzalutamide, or any components of the formulation used.
* Subject has known or suspected brain metastases or active leptomeningeal disease.
* Subject has history of seizure or any condition that may predispose to seizure (e.g., prior stroke or significant brain trauma).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2016-05-08 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (50):
- Belgium (5):
  - Site BE32001, Brussels, Flemish Brabant
  - Site BE32004, Ghent
  - Site BE32007, Hasselt
  - Site BE32003, Kortrijk
  - Site BE32002, Liège
- France (13):
  - Site FR33015, Angers
  - Site FR33009, Caen
  - Site FR33010, Créteil
  - Site FR33014, Le Mans
  - Site FR33013, Lyon
  - Site FR33003, Marseille
  - Site FR33008, Nantes Saint Herblain Cedex
  - Site FR33002, Nîmes
  - Site FR33011, Paris
  - Site FR33001, Paris
  - Site FR33007, Rennes
  - Site FR33005, Suresnes
  - Site FR33012, Villejiuf
- Germany (15):
  - Site DE49005, Nürtingen, Baden-Wurttemberg
  - Site DE49017, Duisburg, North Rhine-Westphalia
  - Site DE49015, Bergisch Gladbach, Northwest
  - Site DE49014, Berlin
  - Site DE49003, Berlin
  - Site DE49009, Bonn
  - Site DE49010, Dresden
  - Site DE49016, Düsseldorf
  - Site DE49004, Göttingen
  - Site DE49001, Hamburg
  - Site DE49008, Hamburg
  - Site DE49007, Hanover
  - Site DE49002, Heidelberg
  - Site DE49012, Münster
  - Site DE49006, Tübingen
- Spain (9):
  - Site ES34004, Santiago de Compostela, A Coruna
  - Site ES34009, Badalona
  - Site ES34011, Barcelona
  - Site ES34006, Barcelona
  - Site ES34008, Barcelona
  - Site ES34001, Madrid
  - Site ES34003, Madrid
  - Site ES34002, Madrid
  - Site ES34010, Madrid
- United Kingdom (8):
  - Site GB44001, Sutton, Surrey
  - Site GB44004, Birmingham
  - Site GB44009, Brighton
  - Site GB44002, Glasgow
  - Site GB44007, London
  - Site GB44003, Northwood, Middlesex
  - Site GB44010, Plymouth
  - Site GB44006, Withington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] de Bono JS, Chowdhury S, Feyerabend S, Elliott T, Grande E, Melhem-Bertrandt A, Baron B, Hirmand M, Werbrouck P, Fizazi K. Antitumour Activity and Safety of Enzalutamide in Patients with Metastatic Castration-resistant Prostate Cancer Previously Treated with Abiraterone Acetate Plus Prednisone for >/=24 weeks in Europe. Eur Urol. 2018 Jul;74(1):37-45. doi: 10.1016/j.eururo.2017.07.035. Epub 2017 Aug 23. PMID 28844372
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=274

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male participants with progressive metastatic castration-resistant prostate cancer were enrolled in this study.
Pre-assignment Details: A total of 272 participants were screened for enrollment & signed an informed consent form, & 57 of those screen failed. The primary reason for screening failure was not fulfilling inclusion/exclusion criteria (52 participants, 19.1%), followed by withdrawal (5 participants, 1.8%).
Period: Overall Study
Arm/Group | Enzalutamide
Started | 215
Treated | 214
Completed | 0
Not Completed | 215
Not completed — Enrolled but Never Received Study Drug | 1
Not completed — Adverse Event | 22
Not completed — Death | 9
Not completed — Progressive Disease | 148
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 8
Not completed — Other: Miscellaneous | 11
Not completed — Lost to Follow-up | 1
Not completed — Other: Transitioned to 9785-CL-0123 | 12

BASELINE CHARACTERISTICS:
Population: The analysis population for all baseline measures consisted of all participants who were enrolled in the study.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — This was an all male study.
  Participants
    Female | 0
    Male | 215
Race/Ethnicity, Customized [Number; unit: Participants] — Race was not collected in France, because of country regulations. Ethnicity was not collected for this study.
  Participants
    White | 165
    Black or African American | 2
    Other | 1
    Not Reported | 47

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Radiographic PFS, was defined as the time from first dose to the first objective evidence of radiographic disease progression or death from any cause, whichever occurred first. For patients with no documented progression event, it was censored on the date of the last disease assessment performed prior to the analysis data cut-off point. Radiographic progression (RP) for soft tissue disease was defined by Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 criteria. RP for bone disease was determined according to the consensus guidelines of a modification of the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) guidelines. The 50th percentile of Kaplan-Meier (KM) estimates was used as the estimate of the rPFS median. A 2-sided 95% Confidence Interval (CI) was provided for this estimate using the Brookmeyer & Crowley (BC) method.
Time Frame: From the first dose of study drug administration up to treatment discontinuation or the data cut-off date of 08 May 2016, whichever occurred first; the median duration of treatment was 5.7 months.
Population: The analysis population consisted of the safety analysis set (SAF) which consisted of all participants who took at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 214
Months | 8.1 [6.11 to 8.28]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose to death from any cause. All events of death were included. If patients discontinued study drug before the analysis data cut-off point, only OS status was assessed every 12 weeks until the data cut-off point date or until death, whichever occurred first. For patients who were alive at the time of the analysis data cut-off point, the OS time was censored on the last date the patient was known to be alive. Death from any cause was included, regardless of whether the event occurred while the patient was still taking study drug or after the patient discontinued study drug. OS median was estimated using the KM method. A 2-sided 95% CI was provided for this estimate using the BC method.
Time Frame: From the first dose of study drug administration up to the data cut-off date of 08 May 2016; up to 2 years.
Population: The analysis population consisted of the SAF.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 214
Months | NA [18.14 to NA] — Could not be estimated due to the low number of events.

3. Secondary Outcome: Percentage of Participants With a Prostate-specific Antigen (PSA) Response
Description: PSA response was defined as at least a 50% decrease from baseline in PSA, and was a binary variable for achieving this criteria (or not) based on the lowest PSA value observed postbaseline. Participants with no postbaseline PSA value were regarded as non-responders. 95% CI for PSA response rate was computed using the Clopper-Pearson method based on the exact binomial distribution.
Time Frame: From the first dose of study drug administration up to the data cut-off date for end-of-study completion 29 Sep 2017; the median duration of treatment was 5.7 months.
Population: The analysis population consisted of the SAF.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 214
Percentage of participants | 22.0 [16.61 to 28.11]

4. Secondary Outcome: Time to PSA Progression
Description: The time to PSA progression was calculated as the time interval from the date of first dose to the date of first observation of PSA progression. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 μg/L (i.e., 2 ng/mL or more) above the nadir or above the baseline value for patients who did not have a decline in PSA postbaseline values, and which was confirmed by a second consecutive value obtained at least 3 or more weeks later (i.e., a confirmed rising trend) (PCWG2 criteria). The 50th percentile of KM estimates was used as the estimate of the time to PSA progression median. A 2-sided 95% CI was provided for this estimate using the BC method.
Time Frame: From the first dose of study drug administration up to the data cut-off date of 08 May 2016; the median duration of treatment was 5.7 months.
Population: The analysis population consisted of the SAF.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 214
Months | 5.7 [5.55 to 5.78]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event occurring or worsening between the start of study treatment date and the latest date of 30 days after the last dose date or the 30-day follow-up visit date, and not later than the data cut-off date or the date of death. AEs, including abnormal clinical laboratory values, were graded using the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) guidelines (V4.03).
Time Frame: From the first dose of study drug administration up to data cut-off date for end-of-study completion (29 Sep 2017); the median duration of treatment was 5.7 months.
Population: The analysis population consisted of the SAF.
Measure: Number; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 214
Participants
  Any TEAE | 199
  NCI-CTCAE Grade ≥3 | 95
  Study Drug-Related | 127
  Study Drug-Related NCI-CTCAE Grade ≥3 | 18
  TEAEs with Death as an Outcome | 22
  Serious Adverse Event (SAE) | 82
  Study Drug-related SAE | 8
  TEAEs Leading to Study Drug Discontinuation | 76
  Study Drug-Related TEAEs Leading to Drug Disc. | 23

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to data cut-off date for end-of-study completion (29 Sep 2017); the median duration of treatment was 5.7 months.
Description: The total number of deaths (all causes) includes deaths reported after the time frame above.
Groups:
- Enzalutamide Total: Participants received 160 mg of enzalutamide orally once daily until they experienced an adverse event, disease progression, started new anti-cancer therapy, withdrew consent, or other protocol-specified criteria.
Arm/Group | Enzalutamide Total
All-Cause Mortality (participants affected / at risk) | 73/214
Serious Adverse Events (participants affected / at risk) | 82/214
Other Adverse Events (participants affected / at risk) | 182/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Total (N=214)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Death (General disorders) | 1 (1)
Device occlusion (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 10 (13)
Inflammation (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Dental fistula (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (4)
Pneumonia (Infections and infestations) | 4 (4)
Pulmonary sepsis (Infections and infestations) | 1 (2)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Monoclonal immunoglobulin present (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (15)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (2)
Loss of consciousness (Nervous system disorders) | 1 (1)
Monoparesis (Nervous system disorders) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 7 (8)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Vertebral artery thrombosis (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Bladder tamponade (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 7 (8)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 5 (8)
Ureteric stenosis (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epiglottic mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Ileostomy closure (Surgical and medical procedures) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Total (N=214)
Anaemia (Blood and lymphatic system disorders) | 23 (36)
Constipation (Gastrointestinal disorders) | 28 (32)
Diarrhoea (Gastrointestinal disorders) | 27 (29)
Nausea (Gastrointestinal disorders) | 32 (38)
Vomiting (Gastrointestinal disorders) | 11 (17)
Asthenia (General disorders) | 38 (51)
Fatigue (General disorders) | 72 (89)
Oedema peripheral (General disorders) | 18 (19)
Weight decreased (Investigations) | 26 (28)
Decreased appetite (Metabolism and nutrition disorders) | 53 (65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (40)
Back pain (Musculoskeletal and connective tissue disorders) | 37 (41)
Bone pain (Musculoskeletal and connective tissue disorders) | 27 (34)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (29)
Dizziness (Nervous system disorders) | 14 (14)
Insomnia (Psychiatric disorders) | 12 (12)
Haematuria (Renal and urinary disorders) | 15 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Hot flush (Vascular disorders) | 12 (12)
Hypertension (Vascular disorders) | 19 (22)

LIMITATIONS AND CAVEATS:
For participants on treatment after the primary analysis data cut-off point (08 May 2016), only AEs were assessed every 24 weeks until treatment discontinuation or death, this was not required for those that enrolled into 9785-CL-0123 (NCT02960022).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.